CLINICAL TRIAL: NCT00513578
Title: Phase 2 Study of Proteinase 3 PR1 Peptide Mixed With Montanide ISA 51 VG Adjuvant and Administered With GM-CSF in Low Risk and Intermediate-1 MDS
Brief Title: Vaccine Therapy and GM-CSF in Treating Patients With Low-Risk or Intermediate-Risk Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Vaccine Company (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000558127; VACCINE-PR1-204
Record Dates: First submitted 2007-08-06; First posted 2007-08-08 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2009-02

CONDITIONS: Myelodysplastic Syndromes
Keywords: refractory anemia with excess blasts; refractory anemia with ringed sideroblasts; refractory anemia; refractory cytopenia with multilineage dysplasia; de novo myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia, Refractory, with Excess of Blasts; Anemia, Refractory | interventions — incomplete Freund's adjuvant; sargramostim

INTERVENTIONS:
Biological: PR1 leukemia peptide vaccine
Biological: incomplete Freund's adjuvant
Biological: sargramostim

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill cancer cells. Colony-stimulating factors, such as GM-CSF, increase the number of white blood cells and platelets found in bone marrow or peripheral blood. Giving vaccine therapy together with GM-CSF may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving vaccine therapy together with GM-CSF works in treating patients with low-risk or intermediate-risk myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the immunologic response, using a PR1-HLA-A2 tetramer assay, to 4 subcutaneous injections of PR1 leukemia peptide vaccine formulated in incomplete Freund's adjuvant (IFA) followed by sargramostim (GM-CSF) in patients with low- and intermediate-1-risk myelodysplastic syndromes.

Secondary

* To determine if non-immunologic responders to 4 subcutaneous injections of PR1 leukemia peptide vaccine formulated in IFA followed by GM-CSF can be converted to immunologic responders by administering 4 additional doses of this treatment.
* To determine the clinical response to 4 or 8 subcutaneous injections of this vaccine.

OUTLINE: This is a multicenter study.

Patients will receive proteinase PR1 leukemia peptide vaccine (TVC-PR1) conjugated with incomplete Freund's adjuvant administered subcutaneously with sargramostim (GM-CSF). Patients will receive a series of four vaccinations at 3-week intervals. Non-immunologic responders after 4 doses of vaccine are eligible to receive 4 additional doses of TVC-PR1 vaccine with the same dose and same dosing intervals. Patients who mount an immunologic response after 4 doses will not receive additional doses of TVC-PR1 vaccine.

After completion of study therapy, patients are followed monthly for up to 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Diagnosis of myelodysplastic syndromes (MDS) and must meet all of the following criteria:

  * FAB class refractory anemia (RA), RA with excess blasts (RAEB), or RA with ringed sideroblasts (RARS)
  * WHO Classification RA, RARS, refractory cytopenia with multilineage dysplasia (RCMD), RCMD with ringed sideroblasts, or RAEB-1
  * Less than 20% blasts on marrow aspirate
  * IPSS risks groups intermediate-1- OR transfusion dependent low-risk
  * Patients with de novo or therapy-related MDS eligible
* HLA-A2 positive at one allele

Exclusion criteria:

* RAEB in transformation or RAEB-2
* Chloroma
* Marrow blasts on aspirate ≥ 20%
* Blood blasts > 1%
* Inaspirable bone marrow
* History or current myelosclerosis occupying > 30% of marrow space
* History of acute myeloid leukemia
* Other causes of cytopenia not related to MDS (i.e., gastrointestinal blood loss)

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0 or 1
* Women of childbearing potential must have a negative serum pregnancy test within 30 days of starting study drug
* Male or female of child-bearing potential must agree to use adequate contraceptive methods
* Serum bilirubin < 2 mg/mL
* Creatinine ≤ 1.5 mg/mL
* ALT < 2 times upper normal limit
* Antineutrophil cytoplasmic antibody (cANCA) negative

Exclusion criteria:

* Pregnant or lactating
* Iron absence on marrow examination or transferrin saturation < 20% and serum ferritin < 50ng/mL
* B12 deficiency
* Folate deficiency
* History of immune-related hematological disorder (i.e., idiopathic thrombocytopenic purpura, autoimmune hemolytic anemia)
* Life expectancy severely limited by diseases other than MDS
* Prior history of malignancy other than MDS (except basal cell or squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for ≥ 5 years
* Known allergy to incomplete Freund's adjuvant
* Hypercalcemia
* Progressive viral or bacterial infection

  * All infections must be resolved and the patient has remained afebrile for seven days without antibiotics
* Cardiac disease of symptomatic nature or cardiac ejection fraction < 40%
* History of Wegener granulomatosis or vasculitis
* Symptomatic pulmonary disease or FEV_1, FVC, and DLCO ≤ 50% predicted
* History of HIV positivity or AIDS
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form or that will place the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret the data

PRIOR CONCURRENT THERAPY:

Exclusion criteria:

* Has received specific therapy for MDS within the past 4 weeks
* Prior allogeneic or syngeneic transplant
* Prior solid organ transplant
* Chronic use (> 2 weeks) of greater than physiologic doses of a corticosteroid agent (dose equivalent to > 10 mg/day of prednisone) within 30 days of the first day of study drug treatment

  * Topical and inhaled corticosteroids are permitted
* Experimental therapy, cyclosporine, antithymocyte globulin, or tacrolimus within 3 months of study entry
* Treatment with androgenic hormones, danazol, colony-stimulating factors, erythropoietin, thalidomide, arsenic trioxide or other agents used to treat MDS within four weeks of the first day of study treatment
* Prior vaccine therapy for MDS
* Prohibited medications during study, including any of the following:

  * Systemic steroids except as required for transfusion reactions
  * Chemotherapy or other investigational drugs
  * Sargramostim (GM-CSF) (except as part of study regimen)
  * Filgrastim (G-CSF)
  * Interleukin-11

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Immunologic response after four injections of vaccine formulation as determined by an increase in the absolute PR1-HLA-A2 tetramer count by at least 0.5/μl

SECONDARY OUTCOMES:
Conversion of non-immunologic responders to immunologic responders by administering 4 additional doses of vaccine
Clinical response as determined by modified IWG criteria

CONTACTS AND LOCATIONS:
Overall Officials: Craig S. Rosenfeld, MD, Study Chair — The Vaccine Company
Locations (1):
- M. D. Anderson Cancer Center at University of Texas, Houston, Texas, United States